CLINICAL TRIAL: NCT04894123
Title: A Phase II Study Evaluating the Rate of Cardiovascular Events During Trifluridine/Tipiracil +/- Oxaliplatin Treatment in Colorectal/Oesogastric Adenocarcinoma Patients That Have Experienced a Past Episode of Thoracic Angina-related Pain Due to Chemotherapy Including 5-fluorouracil/Capecitabine
Brief Title: Cardiovascular Events From Trifluridine/Tipiracil +/- Oxaliplatin in Colorectal/Oesogastric Adenocarcinoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOTAS G-098
Record Dates: First submitted 2021-05-16; First posted 2021-05-20 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Adenocarcinoma; Oesogastric
Keywords: cardiac toxicity
MeSH Terms: conditions — Cardiotoxicity | interventions — trifluridine tipiracil drug combination; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trifluridine/tipiracil +/- oxaliplatin (Experimental): Trifluridine/tipiracil 35 mg/m² orally twice a day from day 1 to day 5 plus oxaliplatin 85 mg/m² intravenous at day 1 every 14 days.
  If oxaliplatin is stopped for neurotoxicity, allergic reaction or other reason, or it is not indicated, patients will continue trifluridine/tipiracil in monotherapy 35 mg/m² orally twice a day between days 1-5 and days 8-12; repeated every 28 days.
  Interventions: Drug: Trifluridine/Tipiracil; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — Trifluridine/tipiracil : 35 mg/m² orally twice a day from day 1 to day 5 every 14 days.
  If oxaliplatin is stopped or it is not indicated, trifluridine/tipiracil in monotherapy 35 mg/m² orally twice a day between days 1-5 and days 8-12; repeated every 28 days.
  Other Names: Lonsurf
Drug: Oxaliplatin — Oxaliplatin : 85 mg/m² intravenous at day 1 every 14 days.
  Other Names: Eloxatin

SUMMARY:
The purpose of this study is to assess the incidence of cardiovascular events in patients with esophageal/stomach or colorectal cancer treated by trifluridine/tipiracil +/- oxaliplatin after an episode of cardiac angina-related thoracic pain due to fluoropyrimidines in the adjuvant or metastatic setting .

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 14-day screening period to determine eligibility for study entry. Patient who meet the eligibility requirement will be included in the study and will be treated by trifluridine/tipiracil +/- oxaliplatin.

ELIGIBILITY:
Inclusion criteria

1. Signed and dated informed consent and willingness to comply with all study procedures and availability for the study duration,
2. Histologically confirmed oesogastric, gastric, colon and/or rectum adenocarcinoma
3. Patients with metastatic non-resectable (oesogastric or colorectal) or adjuvant (colorectal stage III) adenocarcinoma previously treated by fluoropyrimidines (5-FU or capecitabine),
4. Age ≥18 years,
5. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2,
6. Patients who presented an episode of cardiac angina-related thoracic pain due to 5- FU or capecitabine (minimum 21 days [3 weeks] between event and inclusion) at least one of the following events:

   * Instable angina,
   * Acute coronary syndrome (ACS) without ST-segment elevation nor troponin rise.
7. Contraindication to continue treatment with 5FU or capecitabine confirmed and documented by a cardiologist,CONFIDENTIAL Protocol ACOTAS version 1.5, 14/06/2021 Page 32 of 93
8. Indication to receive trifluridine/tipiracil ± oxaliplatin considered better than absence of therapy (colo-rectal stage III) or the best alternative therapy (metastatic colo-rectal and oeso-gastric or gastric) confirmed by a Multidisciplinary Consultation Meeting
9. No contraindication to receive trifluridine/tipiracil (related toxicity),
10. No prior treatment with trifluridine/tipiracil,
11. Following laboratory values obtained within 14 days (2 weeks) prior to start of study treatment:

    * Hematological status: absolute neutrophil count (ANC) ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L; hemoglobin ≥ 9 g/dL,
    * Adequate renal function: serum creatinine level < 150 µM and creatinine clearance ≥ 50 ml/min using the Cockroft-Gault formula,
    * Adequate liver function: serum total bilirubin ≤ 1.5 x upper limit of normal (ULN), alkaline phosphatase (ALP) < 5 x ULN, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN,
12. For female patients of childbearing potential, negative serum pregnancy test within 7 days (1 week) prior starting the study treatment,
13. Female patients of childbearing potential must commit to using reliable and effective methods of contraception during the trial and until at least 12 months after the end of study treatment. Male patients with a partner of childbearing potential must agree to use effective contraception in addition to the contraceptive method used by their partner during the trial and until at least 9 months after the end of study treatment.
14. Registration in a national health care system (PUMa - Protection Universelle Maladie included)

Exclusion Criteria:

1. For metastatic colo-rectal-cancer, MSI and/or dMMR tumor
2. For metastatic oeso-gastric and gastric adenocarcinoma, HER+++ or HER++ FISH positive tumor
3. Left ventricular dysfunction with a left ventricular ejection fraction (LVEF) < 35% with or without an automatic implantable defibrillator,
4. Non-revascularized multivessel coronary artery disease,
5. ACS with ST elevation, and/ or troponin rise
6. QT/QTc interval > 470 ms (for women) and > 450 ms (for men) NB: Caution is required when using medicinal products with human thymidine kinase substrates, e.g. zidovudine and other drugs known to prolong the QTc interval (exhaustive list on https: //www.crediblemeds.org.")
7. Documented coronary vasospasm during 5-FU treatment leading to myocardial infarction,
8. Pregnancy and breastfeeding,
9. Treatment with any other investigational medicinal product within 28 days (4 weeks) before start of the study treatment,
10. Rare hereditary problems of galactose intolerance, the Lapp lactose deficiency, or glucose-galactose malabsorption,
11. Any other serious and uncontrolled non-malignant disease,
12. Major surgery or traumatic injury within 28 days (4 weeks) before the start of study treatment,
13. Patients with known allergy to any excipient to study drugs,
14. Bowel obstruction or inability to swallow tablets,
15. Peripheral neuropathy Grade > 1 for the oxaliplatin schedule,
16. Non resolved non-hematological toxicities from prior therapies (grade >2),
17. Abnormal values at inclusion for :

    * kalemia ;
    * Magnesemia;
    * Calcemia and corrected calcium level
18. Patient under a legal protection regime (guardianship, curatorship, judicial safeguard), or administrative decision, or incapable of giving his/her consent
19. Impossibility of submitting to the medical follow-up of the study for geographical, social reasons or psychiatric illness.
20. Patients admitted to a health or social establishment for purposes other than that of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Rate of cardiovascular events at 3 months. | At 3 months
  Assessment of the rate of cardiovascular events in patients treated by trifluridine/tipiracil +/- oxaliplatin over a 3-month period.

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events by CTCAE 5.0 | Assessed up to 48 months
  Safety profile of the trifluridine/tipiracil and oxaliplatin combination
Number of patients with disease control rate (DCR) | Assessed up to 48 months
  DCR defined as partial response, complete response (CR), or stable disease (SD).
The 3-month drop-out rate of limiting toxicity | At 3 months
  Drop-out rate defined as the number of patients who left the study due to limiting toxicity between treatment initiation and 3 months.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU Jean Minjoz, Besançon
  - Centre Hospitalier Boulogne/ Mer, Boulogne-sur-Mer
  - Hôptial Henri Mondor, Créteil
  - Chu Dijon, Dijon
  - Hôpital Privé Jean Mermoz, Lyon
  - GH Pitié Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
  - CHU Poitiers, Poitiers
  - Hôpital Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - CHU Tours Hôpital Trousseau, Tours

IPD SHARING:
Plan to Share IPD: No